CLINICAL TRIAL: NCT05533983
Title: A Phase II Study of Fecal Microbiota Transplantation With Nivolumab in Patients With Advanced Solid Cancers Who Have Progressed During Anti-PD-(L)1 Therapy
Brief Title: FMT With Nivolumab in Patients With Advanced Solid Cancers Who Have Progressed During Anti-PD-(L)1 Therapy
Acronym: NIVO-FMT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Sook Ryun Park, Associate Professor, Asan Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022-0761
Record Dates: First submitted 2022-09-06; First posted 2022-09-09 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-04

CONDITIONS: Solid Carcinoma
MeSH Terms: interventions — Fecal Microbiota Transplantation; Nivolumab

STUDY DESIGN:
Intervention Model Description: This is a single-center, open-label, Phase 2 study to evaluate the efficacy and safety of FMT with nivolumab in patients with advanced, unresectable, or metastatic solid cancer who have progressed during anti-PD-(L)1 therapy.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Preparation of Frozen Stool Suspensions for FMT (Experimental): The study will enroll patients with advanced, unresectable, or metastatic solid cancer who have progressed during anti-PD-(L)1 therapy.
  Interventions: Other: fecal microbiota transplantation with Nivolumab

INTERVENTIONS:
Other: fecal microbiota transplantation with Nivolumab — This is a single-center, open-label, Phase 2 study to evaluate the efficacy and safety of FMT with nivolumab in patients with advanced, unresectable, or metastatic solid cancer who have progressed during anti-PD-(L)1 therapy.
  Other Names: FMT; Nivolumab

SUMMARY:
This is a single-center, open-label, Phase 2 study to evaluate the efficacy and safety of FMT with nivolumab in patients with advanced, unresectable, or metastatic solid cancer who have progressed during anti-PD-(L)1 therapy.

DETAILED DESCRIPTION:
A single donor-derived FMT will be administered two times in a 2-week interval (± 5 days), which composes one set of FMT. If clinical benefit (complete response [CR], partial response [PR], or stable disease [SD]) is not observed with the 1st set of FMT in the first evaluation of response, the 2nd set of FMT from another donor will be administered unless rapid progression of disease, rapid clinical deterioration, progressive tumor at critical anatomical sites (e.g., cord compression) requiring urgent alternative medical intervention or medical conditions in which further FMT is not the best patient's interest in the opinion of the investigator. If disease progression occurs after achieving clinical benefit (CR, PR, or SD) with the 1st set of FMT, the 2nd set of FMT can be performed using a stool from the same donor as the 1st set of FMT (preferred) or another donor according to the investigator's discretion.

Nivolumab 3 mg/kg iv will be started on day after FMT and followed by additional nivolumab therapy 3 mg/kg iv every 2 weeks until disease progression, intolerable toxicity, or any other of the criteria for treatment discontinuation is met with a maximum of 2-year total duration. In a cycle when FMT is performed, nivolumab will be administered on day after FMT.

ELIGIBILITY:
Donor inclusion criteria Having provided written consent before participation in the study, all donor candidates must fulfil all of the following criteria to be eligible for a donor in this study.

1. Sex: Male or female
2. Age (at the time of informed consent): 19 years and older
3. Subjects with histologically- or cytologically-confirmed solid cancer In case of hepatocellular carcinoma, clinically confirmed diagnosis as per the American Association for the Study of Liver Diseases (AASLD) is allowed.1
4. Patients who currently maintain a CR, PR or SD per RECIST v1.12 for at least 6 months with anti-PD-(L)1 monotherapy for solid cancer

Donor exclusion criteria The subject who meets any of the following criteria will be excluded from a donor candidate. If an enrolled donor candidate is found to meet any of the following criteria anytime during the study, the donated stool obtained when those exclusion criteria are met will not be used for FMT.

1. Having taken antimicrobials (antibiotics, antivirals antifungals) in the 4 weeks prior to donation
2. Positive result for any pathogen tests during the screening period (Table 3)
3. Current gastrointestinal symptoms including diarrhea, nausea, or vomiting
4. History of chronic gastrointestinal disease including inflammatory bowel disease, celiac disease, or irritable bowel syndrome
5. History of systemic autoimmune disease (e.g., multiple sclerosis, connective tissue disorder, type I diabetes mellitus)
6. History of significant neurological (except for chemotherapy-induced neuropathy), neurodegenerative, neurodevelopmental, or psychiatric disorders
7. History or risk behaviors for infectious disease:

   * History of HIV, syphilis, human T-lymphotropic virus I and II
   * Current systemic infection
   * Enteric pathogen infection in the last 8 weeks
   * Vaccination with a live attenuated virus in the last 8 weeks
   * Previous tissue/organ transplant
   * Recent travel (3 months) to tropical countries, countries with endemic diarrheal diseases or high risk of traveler's diarrhea (Africa, Southeast Asia, Mexico, Central America, South America, Caribbean)

Recipient Main Inclusion criteria

Having provided written consent before participation in the study, patients must fulfill all of the following criteria to be eligible for this study:

1. Sex: Male or female
2. Age (at the time of informed consent)L 19 years and older
3. Patients with histologically- or cytologically-confirmed solid cancer In case of hepatocellular carcinoma, clinically confirmed diagnosis as per the American Association for the Study of Liver Diseases (AASLD) is allowed.1
4. Patients who do not have standard treatment, are no longer effective, are not drug resistant to standard treatment, or are unable to use standard treatment, and have previously performed anti-PD-1 or anti-PD-L1-based treatment (as monotherapy or combination therapy)
5. Patients who did not experience any of the following immune-related adverse events (irAEs) during prior immunotherapy:

   * A previous irAE corresponding to treatment discontinuation criteria for nivolumab as described in Section 8.2.2.3
   * Unresolved irAEs prior to study entry (alopecia, Grade ≤2 sensory neuropathy, or other Grade ≤2 AEs not constituting a safety risk based on Investigator's judgment are acceptable)
6. Patients who have at least 1 measurable lesion per the RECIST v1.12 as confirmed by imaging within 28 days before study enrollment. The following requirements should also be satisfied:

   ˙If patients only have lesions that were previously treated with radiation, the lesion should be limited to one with confirmed aggravation by imaging after radiation.
7. Eastern Cooperative Oncology Group (ECOG) performance status score of 0-2
8. Patients with a life expectancy of at least 3 months
9. Patients whose latest laboratory data meet the below criteria within 7 days before the initiation of study treatment. If the date of the laboratory tests at the time of study entry is not within 7 days before the initiation of study treatment, testing must be repeated within 7 days before the initiation of study treatment, and these latest laboratory tests must meet the following criteria. Of note, laboratory data will not be valid if the patient has received a granulocyte colony-stimulating factor (G-CSF) within 7 days before testing.

   * White blood cells ≥2,000/mm3 and neutrophils ≥1,500/mm3
   * Platelets ≥100,000/mm3
   * Hemoglobin ≥9.0 g/dL
   * Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 3.0 x the upper limit of normal (ULN) of the study site (or ≤ 5.0 x ULN of the study site in patients with liver metastases)
   * Total bilirubin ≤ 1.5 x ULN of the study site
   * Creatinine ≤ 1.5 x ULN of the study site or creatinine clearance (either the measured or estimated value using the Cockcroft-Gault equation) > 45 mL/min
10. Women of childbearing potential (including women with chemical menopause or no menstruation for other medical reasons)#1 must agree to use contraception#2 from the time of informed consent until 5 months or more after the last dose of the study treatment. Also, women must agree not to breastfeed from the time of informed consent until 5 months or more after the last dose of the study treatment.
11. Men must agree to use contraception#2 from the start of study treatment until 7 months or more after the last dose of the study treatment.

    * 1. Women of childbearing potential are defined as all women after the onset of menstruation who are not postmenopausal and have not been surgically sterilized (e.g., hysterectomy, bilateral tubal ligation, bilateral oophorectomy). Postmenopause is defined as amenorrhea for ≥12 consecutive months without specific reasons. Women using oral contraceptives, intrauterine devices, or mechanical contraception such as contraceptive barriers are regarded as having childbearing potential.
    * 2. The subject must consent to use any two of the following methods of contraception: vasectomy or condom for patients who are male or female subject's partner and tubal ligation, contraceptive diaphragm, intrauterine device, spermicide, or oral contraceptive for patients who are female or male subject's partner.
12. Patients must be willing to provide blood and fecal samples at baseline, on-treatment, and/or disease progression for biomarker analyses.
13. Patients who have biopsiable lesion(s) must consent to undergo fresh tumor biopsies of accessible lesion(s).

Recipient Main Exclusion criteria Patients who meet any of the following criteria at the time of assessment for study entry will be excluded. If an enrolled subject is found to meet any of the following criteria before the initiation of study treatment, the subject will not be started on study treatment and will be withdrawn from the study.

1. Patients with active malignancy within the previous 2 years before study entry (with the exception of completely resected non-melanoma skin cancer, curatively treated carcinoma in situ or intramucosal carcinoma, superficial bladder cancer treated with curative intent, localized prostate cancer treated with curative intent or other cancers that are less likely to influence on their prognosis such as localized thyroid papillary carcinoma)
2. Patients with residual adverse effects of prior therapy or effects of surgery that would affect the safety evaluation of the study treatment in the opinion of the investigator or sub-investigator.
3. Patients with current or past history of severe hypersensitivity to any other antibody products
4. Patients with active autoimmune disease with systematic treatment (i.e., immunomodulator, corticosteroid, or immunosuppressant) required within the past 2 years before study entry.

   * Replacement therapy (e.g., thyroxine, insulin, or physiological corticosteroid replacement therapy due to dysfunction of adrenal gland or pituitary gland, etc.) is not regarded as a form of systematic treatment and would be allowed.
   * Patients with eczema, psoriasis, lichen simplex chronicus, or vitiligo with dermatologic manifestations only (e.g., no psoriatic arthritis) may be eligible provided that they meet the following conditions:

     * Rash must cover less than 10% of the body surface area.
     * Disease is well controlled at baseline and only requires low potency topical steroids.
5. Patients with a current or past history of interstitial lung disease or pulmonary fibrosis diagnosed based on imaging or clinical findings. Patients with radiation pneumonitis may be enrolled if the radiation pneumonitis has been confirmed as stable (beyond acute phase) without any concerns about recurrence.
6. Patients with concurrent diverticulitis or symptomatic gastrointestinal ulcerative or inflammatory disease (e.g., Crohn´s disease or ulcerative colitis)
7. Patients with any metastasis in the brain or meninx that is symptomatic or requires treatment. Patients may be enrolled if the metastasis is asymptomatic and requires no treatment.
8. Patients with uncontrollable pericardial fluid, pleural effusion, or ascites requiring frequent drainage (recurrence within 2 weeks of intervention)
9. Patients with uncontrollable, tumor-related pain
10. Patients who have experienced a transient ischemic attack or cerebrovascular accident within 180 days before study entry
11. Patients with a history of uncontrollable or significant cardiovascular disease meeting any of the following criteria:

    * Myocardial infarction within 180 days before study entry
    * Uncontrollable angina pectoris within 180 days before study entry
    * New York Heart Association (NYHA) Class III or IV congestive heart failure
    * Uncontrollable hypertension despite appropriate treatment (e.g., systolic blood pressure ≥150 mmHg or diastolic blood pressure ≥ 90 mmHg lasting 24 hours or more)
    * Clinically significant cardiac arrhythmia not controlled by adequate medication
12. Patients receiving or requiring anticoagulation therapy for a disease. Patients receiving antiplatelet therapy including low-dose aspirin may e enrolled.
13. Patients with uncontrollable diabetes mellitus
14. Patients with systemic infections requiring treatment within 14 days before starting the study treatment
15. Patients who have a condition requiring systemic corticosteroids (> 10 mg daily prednisone or equivalents) (except for temporary use, e.g., for examination or prophylaxis of allergic reactions) or other immunosuppressants within 28 days before study entry

    ˙Patients are permitted to use topical, ocular, intra-articular, intranasal, and inhalational corticosteroids (with minimal systemic absorption)
16. Patients who have a history of organ transplant, including stem cell allograft
17. Patients who have received antineoplastic drugs (e.g., chemotherapy agents, molecular-targeted therapy agents, or immunotherapy agents) within 28 days before starting the study treatment, except for anti-PD-(L)1 inhibitor such as nivolumab, pembrolizumab, atezolizumab, avelumab, or durvalumab, for which its regular cycle interval is required before starting the study.
18. Patients who have undergone surgical adhesion of the pleura or pericardium within 28 days before starting the study treatment
19. Patients who have undergone major surgery under general anesthesia within 28 days before starting the study treatment
20. Patients who have received radiotherapy within 28 days before starting the study treatment or radiotherapy to bone metastases within 14 days before starting the study treatment
21. Patients who have received any radiopharmaceuticals (except for examination or diagnostic use of radiopharmaceuticals) within 42 days before the study treatment
22. Patients with known history of Human Immunodeficiency Virus (HIV) infection
23. Patients with active HBV (detectable HBs antigen or HBV DNA) or HCV infection (detectable HCV RNA):

    * For the subject receiving antiviral agents for HBV at screening, if the subject has been treated for > 2 weeks and HBV DNA is <500 IU/mL (or 2,500 copies/mL) prior to study entry, the subject will be allowed to be enrolled in the study. Antiviral agent should be continued for 6 months after study treatment discontinuation.
    * For hepatocellular carcinoma, patients with past or ongoing HCV infection will be eligible for the study.
24. Women who are pregnant or breastfeeding, or possibly pregnant
25. Patients who have received any other unapproved drug (e.g., investigational use of drugs, unapproved combined formulations, or unapproved dosage forms) within 28 days before starting the study treatment
26. Patients who have received a live vaccine within 4 weeks before starting the study treatment
27. Patients judged to be incapable of providing consent for reasons such as concurrent dementia
28. Other patients judged by the investigator or sub-investigator to be inappropriate as subjects of this study

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-03-08 (Actual); Primary Completion 2026-08-19 (Estimated); Study Completion 2026-08-19 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate | 5year
  ˙ To evaluate the anti-tumor activity (objective response rate [ORR]) of fecal microbiota transplantation (FMT) in combination with nivolumab in patients with advanced solid cancers who have progressed on prior anti-PD-(L)1 based therapy (as monotherapy or combination)

CONTACTS AND LOCATIONS:
Overall Officials: Sook Ryun Park, M.D, Ph D, Principal Investigator — Asan Medical Center, Ulsan University of College of Medicine
Locations (1):
- Asan Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No